CLINICAL TRIAL: NCT05991427
Title: A Phase I, Randomized, Observer Blind Clinical Trial to Evaluate the Safety and Immunogenicity of Recombinant Zoster Vaccine (Adenovirus Vector) in Healthy Adults Aged 50-65 Years
Brief Title: A Study to Evaluate the Safety and Immunogenicity of ChAdOx1-VZV in Healthy Adults Aged 50-65 Years
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CanSino Biologics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CTP-CVE-001
Record Dates: First submitted 2023-07-28; First posted 2023-08-14 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Herpes Zoster
Keywords: Varicella zoster virus; Safety; Immunogenicity; Intramuscular injection; Inhalation; Vaccine
MeSH Terms: conditions — Herpes Zoster; Chickenpox; Respiratory Aspiration

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Experimental vaccine group, low dose, Intramuscular injection(IM) (Experimental): 2 doses of ChAdOX1-VZV vaccine (1 × 10^10 vp) on Day 0 and Month 4
  Interventions: Biological: Recombinant Zoster Vaccine (Adenovirus Vector) (ChAdOx1-VZV)
- Control vaccine group, low dose, IM (Active Comparator): 2 doses of Shingrix vaccine (0.5ml) on Day 0 and Month 4
  Interventions: Biological: Zoster Vaccine Recombinant, Adjuvanted (Shingrix)
- Experimental vaccine group, high dose, IM (Experimental): 2 doses of ChAdOX1-VZV vaccine (5 × 10^10 vp) on Day 0 and Month 4
  Interventions: Biological: ChAdOx1-VZV
- Control vaccine group, high dose, IM (Active Comparator): 2 doses of Shingrix vaccine (0.5ml) on Day 0 and Month 4
  Interventions: Biological: Shingrix
- Experimental vaccine group, Aerosol, Inhalation(IH) (Experimental): 2 doses of ChAdOX1-VZV vaccine (2 × 10^10 vp) on Day 0 and Month 4
  Interventions: Biological: IH ChAdOx1-VZV
- Saline group, Aerosol, IH (Placebo Comparator): 2 doses of saline (0.2ml) on Day 0 and Month 4
  Interventions: Biological: IH saline

INTERVENTIONS:
Biological: Recombinant Zoster Vaccine (Adenovirus Vector) (ChAdOx1-VZV) — 2 doses of ChAdOX1-VZV vaccine on Day 0 and Month 4
  Arms: Experimental vaccine group, low dose, Intramuscular injection(IM)
Biological: Zoster Vaccine Recombinant, Adjuvanted (Shingrix) — 2 doses of Shingrix vaccine on Day 0 and Month 4
  Arms: Control vaccine group, low dose, IM
Biological: ChAdOx1-VZV — 2 doses of ChAdOX1-VZV vaccine on Day 0 and Month 4
  Arms: Experimental vaccine group, high dose, IM
Biological: Shingrix — 2 doses of Shingrix vaccine on Day 0 and Month 4
  Arms: Control vaccine group, high dose, IM
Biological: IH ChAdOx1-VZV — 2 doses of ChAdOX1-VZV vaccine on Day 0 and Month 4
  Arms: Experimental vaccine group, Aerosol, Inhalation(IH)
Biological: IH saline — 2 doses of saline on Day 0 and Month 4
  Arms: Saline group, Aerosol, IH

SUMMARY:
This is a randomized, observer blind and controlled study. Participants in low-dose and high-dose IM group will be randomized in a ratio of 2:1 to receive either the investigational product or the control. Participants in the IH group will receive either inhaled investigational product or saline in a ratio of 3:1. Enrollment will be in an ascending order of dosage groups. All participants will receive 2 doses in 4 months interval. Blood samples will be collected for immunogenicity evaluation over the time course of the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants who can understand and comply with the study procedures, understand the risks involved in the study, and provide written informed consent
* Male and female volunteers aged 50 to 65 years at time of informed consent.
* Healthy or in stable health participants with pre-existing, stable, well-controlled disease, defined as mild disease or medical condition not requiring medical therapy or not requiring a change in medical therapy due to worsening of disease during the 6 months before enrollment may be enrolled at the discretion of the investigator.
* Female participants of childbearing potential must have a negative urine pregnancy test at screening and before each dose of investigational vaccine and have been using an adequate form of contraception 30 days prior to first dose of investigational vaccine and agree to use adequate contraception for the entire duration of their participation in the study.
* Male participants must agree to use adequate contraception from the first dose of investigational vaccine until at least 30 days after the last dose of investigational vaccine.

Exclusion Criteria:

* Pregnant or lactating at screening or planning to become pregnant (self or partner) at any time during the study, including the follow-up period
* History of severe allergic reaction (e.g., anaphylaxis) to any component of the vaccine.
* History of herpes zoster (HZ) (Shingles) in the past 5 years.
* Previous vaccination against HZ.
* History of or present substance abuse as judged by the investigator.
* Immunosuppression resulting from hematopoietic stem cell transplantation, acquired immunodeficiency syndrome (AIDS) or symptomatic (human immunodeficiency virus) HIV infection.
* Chronic administration of immunosuppressants (at least 10 mg per day of prednisone equivalent for glucocorticoids) or other immune-modifying drugs within 6 months prior to the first dose of investigational vaccine.
* Has received any blood products or immunoglobulin within 90 days prior to study injection, or is likely to require infusion of blood products during the study period.
* Is undergoing chemotherapy or expected to receive chemotherapy during the study period; has a diagnosis of or receiving treatment for cancer within the last 5 years.
* History of clinically significant thrombocytopenia or other clotting disorders.
* Serious cardiovascular disease (pulmonary heart disease, pulmonary edema, hypertension that cannot be controlled by medication (systolic blood pressure > 160 mmHg and/or diastolic blood pressure > 100 mmHg)), serious liver and kidney disease, and diabetes mellitus with complications.
* History of allergic skin diseases.
* Use of any investigational or non-registered product (drug or vaccine) within 30 days before the first dose of investigational vaccine/product, or planned use during the study period.
* Receipt of any other immunizations within one month before the first dose of investigational vaccine (2 weeks in the case of inactivated influenza vaccines or other non-replicating immunization products [e.g., tetanus and reduced dose diphtheria toxoid (dT) vaccine, pneumococcal vaccine, hepatitis A vaccine, hepatitis B vaccine]), or scheduled within 30 days after last dose of investigational vaccine.
* Received a vaccine with adenovirus vector within 6 months prior to the first dose of investigational vaccine.
* Investigator site staff directly involved in the conduct of the study, site staff otherwise supervised by the investigator, and their respective family members.
* Volunteers with or have history of lung function abnormalities such as asthma, chronic obstructive pulmonary disease, and pulmonary fibrosis.
* Current smokers.
* History or current evidence of any condition, therapy, or laboratory abnormal values that are clinically significant which might confound the results of the study, interfere with the participant's participation for the full duration of the study, or is not in the best interest of the participants to participate, in the opinion of the treating investigator.

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2023-11-07 (Actual); Primary Completion 2024-11-04 (Actual); Study Completion 2024-11-04 (Actual)

PRIMARY OUTCOMES:
Incidence of local and systemic reactogenicity within 7 days after each vaccination | Within 7 days after each vaccination
Incidence of Serious Adverse Event (SAE) and Adverse Event of Special Interest (AESI) from the 1st dose to the end of study. | From the 1st dose to the end of study

SECONDARY OUTCOMES:
The unsolicited adverse events for 28 days after each vaccination | 28 days after each vaccination
The blood biochemistry parameters, include Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST), Basophils (BAS), Creatinine (CREA), Eosinophils (EOS), Fibrinogen (FIBR), Hematocrit (HCT), Hemoglobin (HGB), on day 7 post each vaccination. | Day 7 post each vaccination
The Geometric mean titer (GMT) of gE-specific antibody using Enzyme-linked Immunosorbent Assay (ELISA) over the time course. | Through study completion, an average of 8 months
The GMT of gE-specific antibody 28 days after the 1st and 2nd dose vaccination across each vaccination group. | 28 days after the 1st and 2nd dose vaccination
The gE-specific IFN-γ by EliSpot over the time course of the study | Through study completion, an average of 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Scot Halperin, MD, Principal Investigator — Canadian Center for Vaccinology
Locations (1):
- Canadian Center for Vaccinology, Halifax, Canada